CLINICAL TRIAL: NCT03228160
Title: Effects of Linearly Polarized Near-Infrared Irradiation in Patients With Sympathetically Maintained Neuropathic Pain Syndrome
Brief Title: Light Irradiation and Outcome for Neuropathic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Chun-De Liao, PT, Physical therapist, Taipei Medical University Shuang Ho Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N201511030
Record Dates: First submitted 2016-01-29; First posted 2017-07-24 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Complex Regional Pain Syndrome
Keywords: Sympathetically Maintained Pain; Linear-Polarized Near-Infrared Irradiation; Stellate Ganglion; Heart Rate Variability; Autonomic Dysfunction Outcome
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — Phototherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SGI irradiation (Experimental): Experimental group with active Linearly Polarized Near-Infrared light irradiation to stellate ganglion.
  Interventions: Other: Linearly Polarized Near-Infrared light Irradiation
- Shame irradiation (Sham Comparator): Control group with shame Linearly Polarized Near-Infrared light irradiation to stellate ganglion.
  Interventions: Other: Linearly Polarized Near-Infrared light Irradiation

INTERVENTIONS:
Other: Linearly Polarized Near-Infrared light Irradiation — The SGI was carried out with the use of a linear-polarized near-infrared irradiation device, Minato Alphabeam Infrared Ray Therapy Unit (Minato Medical Science Co., Ltd., Hyogo, Japan), by a senior physical therapist. The maximum output was 3000 mW/cm² at wavelengths of 0.7 to 1.6 m-⁶, including a combination of red and near-infrared radiation. All patients in the experimental group received SGI under the conditions as follows: output, 90%; irradiation circle 1:2 (irradiation 3 seconds followed by 7-seconds pause); duration of irradiation, 10 min; and total irradiation energy density, 194.8 J/cm². The instrument in the control group with shame irradiation was the same as that in the experimental group with the exception that emitted radiation from device was inactive.
  Other Names: Phototherapy

SUMMARY:
Background. Sympathetically maintained pain (SMP) can be effectively relieved by light irradiation to the area near stellate ganglion (SGI), which is applied as an alternative to sympathetic blockade. The clinical efficiency of SGI on heart rate variability (HRV) and its association with pain outcome need to be further identified.

Objectives. This study is aimed to identify the effects of SGI on pain, HRV indices, quality of life, and function outcomes.

Design. A prospective, double blind, randomized designed study Setting. An outpatient pain medicine clinic Subjects and Methods. A total of 44 patients will be enrolled and randomized to their allocations: the experimental group (EG, n=22) and control group (CG, n=22). All patients in EG will receive 12 sessions (twice a week) of standard SGI, while those in CG go through the same protocol except a shame irradiation is applied. Pain, HRV variables, quality of life, and function outcoms are measured before and after SGI in each session. All measures at the first-half and second-half courses are analyzed.

DETAILED DESCRIPTION:
Sympathetically maintained pain (SMP) is defined as an aspect of pain which is maintained or mediated by sympathetic efferent activity including the action of circulating catecholamine and is often linked to the complex regional pain syndrome (CRPS). SMP has been categorized as a subset of neuropathic pain mediated by the underlying mechanism of peripheral sensitization referring to noradrenergic sensitization of peripheral afferent nociceptive fibers and a pathologically sympathetic-sensory coupling interaction between the efferent sympathetic and the afferent system. Besides, SMP is associated with vasomotor and sudomotor dysfunction through either peripheral integerized by an adrenoreceptor stimulated or central organized by sensitization. Therefore, modulation of sympathetic activity either by means of pharmacological analgesics or local sympathetic ganglion blockade may influence the pain course in patients with chronic pain and hyperalgesia that were suspected to be sympathetically maintained.

The pain associated with sympathetic activity can be relieved by blockage of efferent sympathetic nerves to the affected area. Stellate ganglion block (SGB), a local anesthetic blockade of sympathetic ganglia, has been advocated as an early intervention to achieve sympatholysis and its strong evidence had been identified. However, a success of SGB depends on the skilled invasive technique in application and several potential complications may be elucidated. Alternatively, the light irradiation near the stellate ganglion region (SGI) using either low-reactive level laser or linear-polarized near-infrared light irradiation had been used as a noninvasive method for local anesthetic sympathetic blockade. Furthermore, SGI can be safely and conveniently performed in clinical practice even when an anesthetic physician is not available, had been well tolerated by patients, and no thermal injury or side effects were reported by literatures.

SGI had been identified to offer similar effects of SGB for patients with neuropathic pain, including improving blood flow by dilating vessels and reducing pain by directly blocking afferent nociceptive signal traveling via sympathetic pathways. The irradiation effect on heart rate variability (HRV), which is an objectively non-invasive marker of the autonomic nervous system, had not yet been well established. If the pathogenesis of SMP is closely referred to some abnormality in the function of autonomic nerve system (ANS), it is more necessary to measure autonomic activity for validation rather than pain status, local temperature or peripheral blood flow. Whether the relieved pain level after SGI is associated to HRV changes remains unclear. Identifying the relationship between HRV and pain status following SGI allows the clinicians to set a prompt protocol of phototherapy using SGI, and to accurately follow the outcome of autonomic dysfunction in patients with SMP.

The purpose of this study was to demonstrate the sympatholytic and clinical effects of linear polarized near-infrared irradiation applied on stellate ganglion in patients with SMP.

An experimental design with two groups will be used and a double blind, prospective randomized control trial will be conducted at the chronic pain medicine center in the physical medicine and rehabilitation department. Potential patients will be recruited. The enrolled patients will be randomly assigned to the experimental group or the control group (CG) using a table of random numbers. Patients in the experimental group will receive a 6-week standard SGI treatment protocol (12 irradiation sessions), while those in the control group being undergo a sham irradiation during the same period. Both the investigators and the patients will be blinded to the group assignments. All outcome measures will be collected by a trained research assistant at the baseline admission prior to SGI therapy, before and after SGI at each irradiation session, and at the follow up admission immediately after the end of 6-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Patients who age from 20 to 80 years and have a diagnosis of neuropathetic pain will be recruited from the chronic pain center at our hospital.

Exclusion Criteria:

* Patients who meted the following criteria are excluded:

  1. Diagnosis of glioblastoma,
  2. History of heart disease, serious arrhythmia or pacemaker user,
  3. Simmond disease or postpartum hypopituitarism,
  4. Habitual smoking or consumption of stimulant beverages such as tea, coffee, or alcohol, and
  5. Any other condition that is unsuitable for phototherapy by a doctor's evaluation.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale (VAS: 0-100mm) | Baseline
  A visual analogue scale (VAS: 0-100mm) representing pain intensity, where 0 represented no pain and 100 indicated unbearable pain. Participants are instructed to indicate a point on the scale corresponding to the pain intensity. The distance from the left end to the selected point is measured to calculate the pain score in millimeters.
Visual analogue scale (VAS: 0-100mm) | Follow up at 3 months (end of intervention)
  A visual analogue scale (VAS: 0-100mm) representing pain intensity, where 0 represented no pain and 100 indicated unbearable pain. Participants are instructed to indicate a point on the scale corresponding to the pain intensity. The distance from the left end to the selected point is measured to calculate the pain score in millimeters.

SECONDARY OUTCOMES:
Short Form (36) Health Surve (SF-36) | Baseline, follow up at 3 months after end of intervention
  Assessment of quality of life
Short Form (36) Health Surve (SF-36) | Follow up at 3 months after end of intervention
  Assessment of quality of life
Disability of the Arm, Shoulder and Hand (DASH) | Baseline, follow up at 3 months after end of intervention
  Function evaluation of upper quarter
Disability of the Arm, Shoulder and Hand (DASH) | Follow up at 3 months after end of intervention
  Function evaluation of upper quarter
Heart rate variability (HRV) analysis | Baseline, follow up at 3 months after end of intervention
  HRV was measured using an ANSWatch wrist monitor (Taiwan Scientific Co., Taipei, Taiwan).
Heart rate variability (HRV) analysis | Follow up at 3 months after end of intervention
  HRV was measured using an ANSWatch wrist monitor (Taiwan Scientific Co., Taipei, Taiwan).

CONTACTS AND LOCATIONS:
Locations (1):
- Shuang Ho Hospital, Taipei Medical University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No